CLINICAL TRIAL: NCT04191863
Title: PSG in Valproate-induced Nocturnal Enuresis in Children
Brief Title: Sleep Architecture in Valproate-induced Nocturnal Enuresis in Primary School and Preschool Children.
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University Hospital 8
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Epilepsy; Nocturnal Enuresis
Keywords: Valproic acid, enuresis, epilepsy.
MeSH Terms: conditions — Epilepsy; Nocturnal Enuresis; Enuresis | interventions — Valproic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with enuresis: 28 epileptic children with induced secondary nocturnal enuresis in valproate monotherapy.
  Interventions: Other: Clinical, EEG and laboratory assessment at presentation; Drug: Valproate
- Children without enuresis: 232 epileptic children without induced secondary nocturnal enuresis in valproate monotherapy.
  Interventions: Other: Clinical, EEG and laboratory assessment at presentation; Drug: Valproate

INTERVENTIONS:
Other: Clinical, EEG and laboratory assessment at presentation — * The patients' history, clinical, demographic, and laboratory data were acquired.
  * The following tests and imaging studies are routinely done for epilepsy patients receiving valproate treatment and developed nocturnal enuresis, blood urea nitrogen (BUN), serum creatinine (Cr), urinary pH (before and after valproate therapy beginning and at enuresis onset), serum levels and therapeutic doses of valproate.
  * Urinary tract ultrasonography (with full and void bladder).
  * CT brain and EEG.
Drug: Valproate — valproate monotherapy
  Other Names: valprioc acid

SUMMARY:
Our study, retrospectively evaluate the characteristics of and the risk factors for the occurrence of nocturnal enuresis in epileptic children kept on valproate monotherapy.

Epileptic children with the age ranged 5 up to 15 years who were started and kept up on valproate monotherapy. In this study, a child determined to have nocturnal enuresis based on the American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders, fourth edition: "an involuntary voiding of urine during sleep, with a severity of at least twice a week, in children aged 5 years or older, in the absence of congenital or acquired defects of the nervous system."

DETAILED DESCRIPTION:
More than 50 years ago, valproic acid has become established as an effective broad-spectrum antiepileptic drug. It is a drug of choice in children and adult with generalized or focal types of epilepsy, and in generalized convulsive status epilepticus. It is used in migraine prophylaxis, and as a modulator of chemotherapy in cancer treatment. Moreover, valproic acid may have a potential role in neuroprotection in stroke patients and head trauma.

NE is one of the side effects of VPA treatment, and it is generally underdiagnosed or overlooked by clinicians. A comprehensive review study, about the effects of valproic acid, did not mention that nocturnal enuresis as an adverse event of the valproate however; more recent study reported variable incidence of VPA-induced NE is 2.2-24%.

The investigator's study, retrospectively evaluate the characteristics of and the risk factors for the occurrence of nocturnal enuresis in epileptic children kept on valproate monotherapy.

Method Participants The study was conducted on 260 children with epilepsy receiving valproate monotherapy aged 5-15 years who attended the outpatient clinic of neurology departments, Mansoura University Hospital, Egypt during the period Sep 2019 to Aug 2019.

Clinical, EEG and laboratory assessment at presentation

* The patients' history, clinical, demographic, and laboratory data were acquired.
* The following tests and imaging studies are routinely done for epilepsy patients receiving valproate treatment and developed nocturnal enuresis, blood urea nitrogen (BUN), serum creatinine (Cr), urinary pH (before and after valproate therapy beginning and at enuresis onset), serum levels and therapeutic doses of valproate.
* Urinary tract ultrasonography (with full and void bladder).
* CT brain and EEG.
* Patients were therefore assessed month to month for a follow up over a time of 6 sequential months, with extra visits as required dependent on seizure recurrence or side effects.

Follow-up at least monthly interval for 6 month for the children kept on valproate monotherapy. Evaluation of seizure control and the reported side effects associated with valproate by the parents were determined. In this way special consideration and directly asking parents about the incidence of NE and its recurrence (daily and monthly) is mandatory.

The time from the initiation of valproate monotherapy to the beginning of NE, the daily dose and the duration of treatment of valproic acid (mg/kg) at the onset of enuresis and the serum level of valproate were reported. Also, the time of cessation of NE either spontaneous or following discontinuation of valproate was determined.

Statistical analysis

A multivariate logistic regression analysis was carried out for the following independent variables: age, weight, body weight, duration of treatment and daily dose of valproate, and serum level valproate. P-value <0.05 were considered of statistically significant results.

ELIGIBILITY:
Inclusion Criteria:

* Epileptic children kept up on valproate monotherapy and developed nocturnal enuresis.
* Age ranged 5 up to 15 years.

Exclusion Criteria:

* Combined therapy with other antiepileptic drugs,
* Abnormal cerebral imaging,
* Poor seizure control,
* Primary nocturnal enuresis (a child didn't accomplish any times of evening dryness -over a time of 6 successive months).
* Congenital or acquired defects of the nervous system.
* Urinary system anomalies, or
* Intellectual disability.

Ages: 5 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: The study was conducted on 260 children with epilepsy receiving valproate monotherapy aged 5-15 years who attended the outpatient clinic of neurology departments, Mansoura University Hospital, Egypt during the period Sep 2019 to Aug 2019.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Nocturnal enuresis | 6 months
  Follow-up at least monthly interval for 6 month for the children kept on valproate monotherapy. The incidence of nocturnal enuresis and its frequency were reported

SECONDARY OUTCOMES:
Side effects of valproic acid | 6 month
  The incidence of the side effects that happened in children during treatment by valproate.

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clayton-Smith J, Bromley R, Dean J, Journel H, Odent S, Wood A, Williams J, Cuthbert V, Hackett L, Aslam N, Malm H, James G, Westbom L, Day R, Ladusans E, Jackson A, Bruce I, Walker R, Sidhu S, Dyer C, Ashworth J, Hindley D, Diaz GA, Rawson M, Turnpenny P. Diagnosis and management of individuals with Fetal Valproate Spectrum Disorder; a consensus statement from the European Reference Network for Congenital Malformations and Intellectual Disability. Orphanet J Rare Dis. 2019 Jul 19;14(1):180. doi: 10.1186/s13023-019-1064-y. PMID 31324220
- [Background] Tomson T, Battino D, Perucca E. Valproic acid after five decades of use in epilepsy: time to reconsider the indications of a time-honoured drug. Lancet Neurol. 2016 Feb;15(2):210-218. doi: 10.1016/S1474-4422(15)00314-2. Epub 2015 Dec 5. PMID 26655849
- [Background] Glauser T, Shinnar S, Gloss D, Alldredge B, Arya R, Bainbridge J, Bare M, Bleck T, Dodson WE, Garrity L, Jagoda A, Lowenstein D, Pellock J, Riviello J, Sloan E, Treiman DM. Evidence-Based Guideline: Treatment of Convulsive Status Epilepticus in Children and Adults: Report of the Guideline Committee of the American Epilepsy Society. Epilepsy Curr. 2016 Jan-Feb;16(1):48-61. doi: 10.5698/1535-7597-16.1.48. PMID 26900382
- [Background] Romoli M, Mazzocchetti P, D'Alonzo R, Siliquini S, Rinaldi VE, Verrotti A, Calabresi P, Costa C. Valproic Acid and Epilepsy: From Molecular Mechanisms to Clinical Evidences. Curr Neuropharmacol. 2019;17(10):926-946. doi: 10.2174/1570159X17666181227165722. PMID 30592252
- [Background] Cattaneo CI, Ressico F, Valsesia R, D'Innella P, Ballabio M, Fornaro M. Sudden valproate-induced hyperammonemia managed with L-carnitine in a medically healthy bipolar patient: Essential review of the literature and case report. Medicine (Baltimore). 2017 Sep;96(39):e8117. doi: 10.1097/MD.0000000000008117. PMID 28953637
- [Background] Badv R S, Abbasi A, Ashrafi M R, Shariatmadari F, Bayat O. The Effect of Sodium Valproate on Urinary Frequency and Enuresis Compared to Carbamazepine in Children with Epilepsy, Iran J Pediatr. 2018 ; 28(6):e66083. doi: 10.5812/ijp.66083.
- [Background] Alshahrani A, Selim M, Abbas M. Prevalence of nocturnal enuresis among children in Primary Health Care Centers of Family and Community Medicine, PSMMC, Riyadh City, KSA. J Family Med Prim Care. 2018 Sep-Oct;7(5):937-941. doi: 10.4103/jfmpc.jfmpc_32_18. PMID 30598936
- [Background] Hamed A, Yousf F, Hussein MM. Prevalence of nocturnal enuresis and related risk factors in school-age children in Egypt: an epidemiological study. World J Urol. 2017 Mar;35(3):459-465. doi: 10.1007/s00345-016-1879-2. Epub 2016 Jun 15. PMID 27306687
- [Background] Kanemura H, Sano F, Ohyama T, Sugita K, Aihara M. The relationship between nocturnal enuresis and sequential changes of NAG/morning urine gravity in epileptic children treated with valproate sodium. J Pediatr Epilepsy 2015;4:61-6.
- [Background] Yamak WR, Hmaimess G, Makke Y, Sabbagh S, Arabi M, Beydoun A, Nasreddine W. Valproate-induced enuresis: a prospective study. Dev Med Child Neurol. 2015 Aug;57(8):737-41. doi: 10.1111/dmcn.12737. Epub 2015 Mar 25. PMID 25808512
- [Background] Fritz G, Rockney R, Bernet W, Arnold V, Beitchman J, Benson RS, Bukstein O, Kinlan J, McClellan J, Rue D, Shaw JA, Stock S, Kroeger Ptakowski K; Work Group on Quality Issues; AACAP. Practice parameter for the assessment and treatment of children and adolescents with enuresis. J Am Acad Child Adolesc Psychiatry. 2004 Dec;43(12):1540-50. doi: 10.1097/01.chi.0000142196.41215.cc. PMID 15564822
- [Derived] Esmael A, Elsherief M, Abdelsalam M, Bendary L, Egila H. Sleep Architecture in Valproate-Induced Nocturnal Enuresis in Primary School and Preschool Children. J Child Neurol. 2020 Dec;35(14):975-982. doi: 10.1177/0883073820944051. Epub 2020 Aug 7. PMID 32762394